CLINICAL TRIAL: NCT02811003
Title: Evaluation of the Rotation Medical Bioinductive Implant for Insertional Achilles Tendinopathy
Brief Title: Achilles Tendon Repair With Bioinductive Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3672-01
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2019-03

CONDITIONS: Tendinopathy
Keywords: Insertional Achilles
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment with Rotation Medical Bioinductive Implant
  Interventions: Device: Rotation Medical Bioinductive Implant

INTERVENTIONS:
Device: Rotation Medical Bioinductive Implant — Placement of bioinductive implant over repair of insertional Achilles tendinopathy

SUMMARY:
To evaluate bioinduction of new tissue and tendon healing after implantation of the Rotation Medical Bioinductive Implant used as adjunct to surgical repair in the treatment of insertional Achilles tendonitis.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm study conducted under a common protocol designed to evaluate long-term outcomes following open treatment and implantation of the Rotation Medical Bioinductive Implant to treat insertional Achilles tendinopathy.

Up to 20 subjects will be enrolled and treated with the Rotation Medical Bioinductive Implant.

Enrollment is anticipated to take up to 12 months and all subjects will be followed for two years after surgery. Therefore, the overall study duration is estimated to be 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age
2. Insertional Achilles tendonitis requiring surgery that has failed conservative management, which consist of:

   A. Shoe modification B. Nonsteroidal anti-inflammatory drugs C. Physical Therapy with/without modalities
3. Chronic Achilles tendon pain lasting longer than 3 months
4. MRI or X-ray of the ankle within 60 days prior to the study procedure
5. Willing to comply with the prescribed post-operative rehabilitation program
6. Willing to be available for each protocol-required follow-up examination
7. Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures
8. Ability to read, understand, and complete subject-reported outcomes in English

Exclusion Criteria:

1. Achilles tendon rupture
2. Previous Achilles tendon surgery on the index ankle
3. Genetic collagen disease
4. History of auto-immune or immunodeficiency disorders
5. History of chronic inflammatory disorders
6. Oral steroid use in last 2 months or injectable steroid use in last 4 weeks
7. History of heavy smoking (> 1 pack per day) within last 6 months
8. Hypersensitivity to bovine-derived materials
9. Hypersensitivity to Polylactic Acid (PLA) and Polyetheretherketone (PEEK) materials
10. Metal implants, fillings, shrapnel, and/or screws
11. Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study
12. Currently involved in any injury litigation or worker's compensation claims relating to the index ankle
13. Enrolled, or plans to enroll, in another clinical trial during this study that would affect the outcomes of this study
14. History of non-compliance with medical treatment, physical therapy/rehabilitation, or clinical study participation
15. History of cognitive or mental health status that interferes with study participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Guyton, MD, Principal Investigator — MedStar Union Memorial Hospital
Locations (2):
- United States (2):
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Allegheny Health Network, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were a total of 20 participants enrolled in the study. The first participant was implanted on 7 June 2016 and the final participant was implanted on 11 August 2017. All participants who were consented and who proceeded to surgery were successfully implanted.
Period: Overall Study
Arm/Group | Treatment
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.60 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17
  African American | 3
Region of Enrollment [Number; unit: participants]
  United States | 20
Height [Mean (Standard Deviation); unit: inches] | 68.30 (4.50)
Weight [Mean (Standard Deviation); unit: pounds (lb)] | 213.30 (38.58)
Study ankle [Count of Participants; unit: Participants]
  Left | 10
  Right | 10
Smoking history [Count of Participants; unit: Participants]
  Never | 14
  Former | 5
  Current | 1
Duration of Achilles pain [Mean (Standard Deviation); unit: months] | 18.10 (11.92)

OUTCOME MEASURES:

1. Primary Outcome: New Tissue Thickness
Description: Measurement of new tissue thickness in millimeters will be made from sagittal magnetic resonance imaging (MRI) at the level of the bone anchor. These measurements were made distal to the attachment of the Achilles tendon, which do not include the thickness of the repaired tendon; therefore, these thicknesses represent the thickness of the newly induced tissue only.
Time Frame: 3, 12, and 24 months
Population: The 3-month MRI for 1 participant did not include the necessary images for thickness measurement; thus, there were only 18 measurements at 3 months. The 12-month MRIs for 3 participants did not include the necessary images for thickness measurement, therefore, there were only 13 measurements at 12 months. The 24-month MRIs for 1 participant did not include the necessary images for thickness measurement, therefore, there were only 15 measurements at 24 months.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Treatment
Number analyzed (Participants) | 18
millimeters
  3 months | 5.40 (1.08)
  12 months: number analyzed (Participants) | 13
  12 months | 5.70 (0.78)
  24 months: number analyzed (Participants) | 15
  24 months | 5.50 (0.92)

2. Primary Outcome: MRI Measurements of Tendon Thickening (Combined Tendon and New Tissue)
Description: Combined measurement of tendon and new tissue thickness in millimeters will be made from sagittal magnetic resonance imaging (MRI) at the insertion (approximately 5-10mm proximal to the bone anchor).
Time Frame: 3, 12, and 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Treatment
Number analyzed (Participants) | 18
millimeters
  3 months | 8.20 (2.47)
  12 months: number analyzed (Participants) | 13
  12 months | 16.80 (4.58)
  24 months: number analyzed (Participants) | 15
  24 months | 18.40 (2.84)

3. Primary Outcome: Tear Rate
Description: Tear rate in the deep portion of the repair at the calcaneus following Achilles surgery will be assessed at each follow-up visit using magnetic resonance imaging (MRI).
Time Frame: following surgery to end of treatment at 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants
  No Tear | 17
  Tear | 3

4. Secondary Outcome: Device Implant Time
Description: Time in minutes from introduction of the bioinductive implant into the surgical field to completion of the last staple
Time Frame: Intraoperatively, up to 9 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment
Number analyzed (Participants) | 20
minutes | 5.40 (1.57)

5. Secondary Outcome: Number of Participants With Procedure Technical Success
Description: The number of participants where the device was successfully delivered and affixed to target tendon location (i.e., study device was successfully implanted).
Time Frame: Intraoperatively, up to 9 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 20
Participants
  Device Successfully Implanted | 20
  Device Not Successfully Implanted | 0

6. Secondary Outcome: CAM Boot Time
Description: Cumulative number of days spent in a controlled ankle motion walking boot (CAM boot).
Time Frame: 1 week following surgery to 12 months
Population: The calculated mean time wearing the boot was based on only 16 patients because 3 patients who wore the boot more than 90 days did not report the actual date they stopped wearing the boot; therefore, the actual time wearing the boot was greater than the calculated mean.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 16
days | 76.30 (29.32)

7. Secondary Outcome: Rehabilitation Visits
Description: Rehabilitation measured by the cumulative number of completed rehabilitation or physical therapy (PT) visits to treat index Achilles.
Time Frame: 4 weeks following surgery to end of treatment at 24 months
Population: Overall number of participants analyzed indicates participants that provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Treatment
Number analyzed (Participants) | 10
visits | 17.90 (8.33)

8. Secondary Outcome: Time to Recovery
Description: Recovery will be measured by days to return to normal daily activity (i.e. full, unrestricted activity).
Time Frame: following surgery to end of treatment at 24 months
Population: Overall number of participants analyzed indicates participants that provided data for this outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 10
days | 167.80 (68.04)

9. Secondary Outcome: Participant Satisfaction
Description: Participant Satisfaction will determined based on the response to the statement "I am satisfied with the results of my surgery." The response will be assessed with a 5-point Likert scale, which has 1 - very dissatisfied, 2 - dissatisfied, 3 - neither satisfied nor dissatisfied, 4 - satisfied, 5 - very satisfied
Time Frame: 12 months
Population: Overall number of participants analyzed that provided data for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 17
Participants
  Very dissatisfied | 1
  Dissatisfied | 1
  Neither satisfied nor dissatisfied | 1
  Satisfied | 7
  Very satisfied | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of surgery through 24 month follow-up.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Muscle, tendon and ligament injury (Injury, poisoning and procedural complications) | 1 (1) — Not related to study device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=20)
Numbness (Nervous system disorders) | 1 (2) — Not related to study device
Inversion Injury (Injury, poisoning and procedural complications) | 1 (1) — Not related to study device
Diabetes (Metabolism and nutrition disorders) | 1 (1) — Not related to study device
Pacemaker Implanted (Surgical and medical procedures) | 1 (1) — Not related to study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT02811003/Prot_SAP_000.pdf